CLINICAL TRIAL: NCT02048709
Title: A Phase I Study of GDC-0919 for Adult Patients With Recurrent Advanced Solid Tumors
Brief Title: Indoleamine 2,3-Dioxygenase (IDO) Inhibitor in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GO29753; NLG9191 (Other: clinicaltrials.gov)
Record Dates: First submitted 2014-01-10; First posted 2014-01-29 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Solid Tumor
MeSH Terms: interventions — navoximod

ARMS (1):
- GDC-0919 Dose Escalation (Experimental): GDC-0919 to be given on an outpatient basis as a single agent. Starting dose of GDC-0919 will be 50 mg by mouth every 12 hour. Patients will receive the study drug daily for 21 days followed by 7 days off for a cycle length of 28 days; or on 28 consecutive days of a 28-day cycle
  Interventions: Drug: GDC-0919

INTERVENTIONS:
Drug: GDC-0919 — Supplied in 50 mg and 200 mg capsules. To be taken every 12 hours with water by mouth on an empty stomach (no food or drink other than water for 2 hours prior to dose). Taken twice daily for 21 days each cycle, followed by 7 days off; or taken twice daily on 28 consecutive days of a 28-day cycle

SUMMARY:
This is an open-label Phase I study to evaluate the safety, tolerability, and pharmacokinetics of escalating oral doses of GDC-0919, an investigational agent intended to inhibit the indoleamine 2,3-dioxygenase 1 (IDO1) enzyme and help the human immune system attack solid tumor cells more effectively.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed solid tumor that is relapsed/refractory to standard therapies or for which no approved or curative therapy exists
* Age > or = 18
* Eastern Cooperative Oncology Group (ECOG) performance status < 2
* Life expectancy > or = 12 weeks
* Adequate hematologic and organ function before initiation of GDC-0919
* For some patients only: Accessible lesions amenable to paired fresh tumor biopsies

Exclusion Criteria:

* Some prior cancer immunotherapies
* Untreated brain metastases
* Active or history of autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with dose-limiting toxicities | 28 days
Number of dose-limiting toxicities | 28 days
Percentage of patients with adverse events | approximately 15 months

SECONDARY OUTCOMES:
Pharmacokinetics: Serum concentrations (Cmax/Steady State) | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Georgia Regents University, Augusta, Georgia, United States

REFERENCES:
- [Derived] Nayak-Kapoor A, Hao Z, Sadek R, Dobbins R, Marshall L, Vahanian NN, Jay Ramsey W, Kennedy E, Mautino MR, Link CJ, Lin RS, Royer-Joo S, Liang X, Salphati L, Morrissey KM, Mahrus S, McCall B, Pirzkall A, Munn DH, Janik JE, Khleif SN. Phase Ia study of the indoleamine 2,3-dioxygenase 1 (IDO1) inhibitor navoximod (GDC-0919) in patients with recurrent advanced solid tumors. J Immunother Cancer. 2018 Jun 20;6(1):61. doi: 10.1186/s40425-018-0351-9. PMID 29921320